CLINICAL TRIAL: NCT00582660
Title: Randomized, Placebo-Controlled, Phase 2B Evaluation of Cyclooxygenase-2 Activity in Surgically Resected Primary Colorectal Adenomas and Carcinomas After 7 Days Pretreatment With Celecoxib
Brief Title: Evaluation of Surgically Resected Colorectal Adenomas and Carcinomas After 7 Days Pretreatment With Celecoxib
Acronym: UAB0040
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pfizer (Industry); Pharmacia (Industry)
Responsible Party: Principal Investigator, Marty Heslin, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F001228004; NQ8-00-02-008 (Other: Pfizer Tracking Number)
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Adenoma; Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Celecoxib; Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study drug BID for 7 days before surgery (Active Comparator): 400 mg Celecoxib the study drug will be given for 7 days before surgery
  Interventions: Drug: Celecoxib
- Placebo for 7 days before surgery (Placebo Comparator): Placebo in a one to one randomization prior to surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — 400 mg twice a day for 7 days prior to surgery
  Other Names: study drug
  Arms: study drug BID for 7 days before surgery
Drug: Placebo — one tablet of placebo will be given for 7 days prior to surgery
  Arms: Placebo for 7 days before surgery

SUMMARY:
The purpose of this study is to assess how effective celecoxib is in limiting production of a hormone, prostaglandin, in the subject's body. It is felt that this hormone is involved in the evolution of pre-cancerous growths in the colon to cancerous stage or in the progression of an existing cancer. To answer this question, some subjects are given the new investigational drug, and other subjects a placebo. A placebo is a capsule that contains inactive ingredients. Only by comparing the response of two subject groups, one receiving placebo (inactive), and one receiving celecoxib (active), will we be able to know whether or not celecoxib actually works. The outcome we are assessing is the hormone activity before and after celecoxib is given.

DETAILED DESCRIPTION:
We propose to test the hypothesis that celecoxib, a specific inhibitor of cyclooxygenase -2 (COX-2), will effectively inhibit the enzymatic activity in all tissues sampled after oral administration of celecoxib for 7 days preoperatively. One hundred twenty patients (120) undergoing standard surgical resection for the treatment of primary colorectal adenomas or carcinomas would be randomized to celecoxib or placebo given for 7 days prior to operation. Peripheral blood will be drawn prior to drug or placebo administration, and then morning of operation. At the time of definitive resection of the specimen, normal intestinal mucosa and primary tumor would be harvested and immediately snap frozen at -80 degrees. Levels of COX-2 activity (prostaglandin production) as well as expression of COX-2 and other markers (matrix metalloproteinases(MMPs), tissue inhibitors of MMPs (TIMPs), cell adhesion and cell cycle control molecules will be evaluated in normal mucosa and primary tumor compared between celecoxib and placebo treated patients.

ELIGIBILITY:
Inclusion criteria:

1. Mass suspicious for carcinoma, clinical diagnosis of adenocarcinoma of the colon (to be histologically confirmed upon study entry) or an adenoma that is not removable by endoscopy.
2. Patient must be undergoing colo-rectal resection
3. age > 18yrs
4. Karnofsky performance status(KPS) > 60.
5. Signed and dated informed consent.
6. Complete history and physical examination within 30 days of study entry.
7. Laboratory evaluations within 30 days of study entry to include: Complete Blood Count(CBC) with differential and platelets, Blood Urea Nitrogen(BUN), creatinine, bilirubin, serum glutamic-oxaloacetic transaminase (SGOT), serum glutamic-pyruvic transaminase(SGPT), lactate dehydrogenase(LDH), alkaline phosphatase, total protein, albumin and carcinoembryonic antigen(CEA).
8. Chest x-ray within 30 days of study entry.
9. The subject has no other serious medical illness, other than that treated by this study, which would limit the ability of the patient to receive protocol therapy, or psychiatric condition which would prevent informed consent.

Absolute exclusion criteria:

1. severe infection ;White Blood Cell Count(WBC) > 2 times normal, fever, sepsis)
2. immunosuppression (steroids, transplant patient)
3. emergent operation(perforation, obstruction).
4. Patients with serum bilirubin or creatinine levels greater than two times the normal upper limit would be excluded.
5. Pregnant or lactating women or subjects of child bearing age who do not practice effective means of birth control
6. Sulfonamide allergy
7. Recurrent or previous history of known ischemic heart disease or thrombotic events as well as any angioplasty or cardiac by-pass procedures in the previous 12 months.

Relative exclusion criteria:

1. Medications taken by the patient that are listed in section 9.0 of this protocol would be reviewed by the enlisting physician prior to entry into the study. Warfarin, aspirin and methotrexate would be stopped prior to protocol entry as these are stopped prior to any surgery. The most common of the listed medications would be ACE inhibitors and furosemide. The dose, schedule and indications of the medications would be reviewed with the patient and a decision regarding entry into the study would be made by the enlisting physician. Other less common medications will be similarly reviewed, however most had little or no clinical side effects despite potential biochemical interactions.
2. Medications known to be COX inhibitors would have to be stopped prior to entry into the study. This would include any aspirin,nonsteroidal antiinflammatory drugs(NSAID) (ibuprofen, naproxen, rofecoxib, celecoxib, Mobic, etc) or over the counter cold medication that might contain these substances. A list of common over-the-counter medications that might contain such substances will be reviewed with the patient and if there are any questions after the study has begun, instructions to call before taking any medications will be given.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J Heslin, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Celecoxib: 400 mg BID given for 7 days before surgery
- Placebo: 1 tablet BID given for 7 days before surgery
Period: Overall Study
Arm/Group | Celecoxib | Placebo
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (1) | 62 (1) | 62 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 14 | 16 | 30
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Witha Change (IMPROVEMENT) in Colo-rectal Adenocarcinoma as Measured by Cyclooxygenase-2 Activity After 7 Days of Celecoxib
Description: The Colo-Rectal adenocarcinoma will be measured by cyclooxygenase-2(COX-2) activity at 7 days post baseline. Cox-2 activity is measured by assessing tumors and normal tissue using "Electron microscope and Tandem mass Spectrometry" methodology though the UAB shared Mass Spectrometry facility. Improvement was measured by 2-fold increase in COX-2 activity from baseline. The methodology used was High Performance Liquid Chromatography(HPLC). additional studies include expression of genes thought to be important in colorectal carcinogenesis: COX-1 and 2, MMP, 2 7, and 9, tissue inhibitor of metalloproteinases(TIMPs) 1 ans 2 and beta-catenin.
Time Frame: baseline to 7 days
Measure: Number; unit: Participant
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 20 | 20
Participant | 2.0 | 2.0

2. Primary Outcome: Subjects With Positive Response 72 Hours After Administration of Study Treatment as Measured by Immunoblot
Description: At 72 hours after start of treatment, the number of subjects with immunoblot demonstrated a 1.5 to 2 fold increase in 15-LOX-1 protein expression in human colorectal adenocarcinoma cell line with epithelial morphology(HT-29) and dihydrolipoamide dehydrogenase(DLD)-1 cells.
Time Frame: baseline to 72 hours
Measure: Number; unit: Participants
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 20 | 20
Participants | 3.0 (0.5) | 0 (0.5)

ADVERSE EVENTS:
Time Frame: From baseline visit to 36 months
Arm/Group | Celecoxib | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
The most prominent factor that limited enrollment was this period of time was at the point that the FDA released its finding about the possible cardiac risks associated with Rofecoxib (VIOXX).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No